CLINICAL TRIAL: NCT06052644
Title: Assessing Cognitive and Health Improvements in the Elderly Via Exercise (ACHIEVE) Study - Optimal Exercise Dose-Response to Enhance Cognition and Physical Condition in Cognitively Impaired Older Adults.
Brief Title: Assessing Cognitive and Health Improvements in the Elderly Via Exercise (ACHIEVE) - Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén-
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Aging; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: To allocate participants to their respective groups, we will employ random sampling facilitated by the Epidat program. This grouping process will remain concealed, ensuring that the individuals responsible for enrolling patients into the intervention phase remain unaware of the group assignments. An independent researcher, uninvolved in the subsequent stages of assessment, intervention, data collection, or database creation, will perform this allocation in advance. The group assignments will be communicated via sealed and completely opaque envelopes. The subsequent analysis of the results will be conducted by a separate researcher who has no involvement in either the group assignment process or the intervention itself.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (CG) (No Intervention): The control group will not carry out any type of intervention. You will receive physical activity recommendations from the Pan American Health Organization, developed by sports science professionals.
- EXPERIMENTAL GROUP 1 (EG1) (Experimental): This group will engage in high-intensity physical exercise for 150 minutes per week, three days a week, with each session lasting 50 minutes. The session structure will include a 5-minute warm-up, 40 minutes of the core phase, and 5 minutes of cool down.
  Interventions: Other: Exercise Dose-Response
- EXPERIMENTAL GROUP 2 (EG2) (Experimental): Participants in this group will perform high-intensity exercise twice a week, with each session lasting 30 minutes. The session structure will include a 5-minute warm-up, 20 minutes of the core phase, and 5 minutes of cool down.
  Interventions: Other: Exercise Dose-Response
- EXPERIMENTAL GROUP 3 (EG3) (Experimental): This group will engage in high-intensity exercise four times a week, with each session lasting 50 minutes. The session structure will include a 5-minute warm-up, 40 minutes of the core phase, and 5 minutes of cool down.
  Interventions: Other: Exercise Dose-Response

INTERVENTIONS:
Other: Exercise Dose-Response — The intervention will last for 12 weeks. Depending on the group, participants will engage in the intervention either four times a week or only two times, with the duration ranging from 30 to 60 minutes per session. Each session will consist of three phases: an initial warm-up phase, a central phase, and a cool-down phase.
  The warm-up phase will focus on joint mobility, beginning with flexion-extension, rotation, and lateral neck flexion while maintaining eye contact with a fixed point. This will be followed by trunk mobility exercises, including rotations.
  The central phase will consist of aerobic and strength training performed at an intensity of 80-85% of the maximum heart rate. Each exercise will be performed intensely for 20 to 30 seconds, followed by a rest period of 10 to 15 seconds before repeating the exercise.
  Arms: EXPERIMENTAL GROUP 1 (EG1); EXPERIMENTAL GROUP 2 (EG2); EXPERIMENTAL GROUP 3 (EG3)

SUMMARY:
In Colombia, a demographic transition is occurring that is reflected in an inverted population pyramid, with an increase in the proportion of older adults due to a better quality of life, as well as a decrease in the young population due to the low birth rate. These changes pose challenges for the healthcare system due to aging and its negative consequences for the body. The rate of aging has increased fourfold since 1950, which means a significant increase in the population of older adults compared to those under 15 years of age. Although exercise has been proven to have positive effects on the physical and cognitive health of older adults, there are still gaps in the literature concerning cognitive impairment in older adults, and the optimal dose to achieve maximum therapeutic potential has not been determined.

Therefore, the purpose of this research is to establish the optimal dose-response relationship to high-intensity exercise for improving cognition in older adults with mild cognitive impairment. A Randomized Controlled Clinical Trial with four groups will be conducted. One of the groups will serve as the control and will not receive treatment, focusing on occupational activities. The other three groups will be experimental, and the frequency and duration of exercise will be modified based on the World Health Organization (WHO) guidelines and a previous systematic research with meta-analysis. In the first experimental group (EG1), the WHO recommendations will be applied, consisting of 150 minutes of high-intensity exercise three times a week in sessions of 50 minutes each. In EG2, participants will perform high-intensity exercise twice a week, with a duration of 30 minutes per session. In EG3, high-intensity exercise will be performed four times per week in sessions of 50 minutes each. All experimental groups will receive high-intensity physical exercise interventions that combine aerobic and strength exercises adapted to the population. The sessions will be divided into three phases: warm-up, core phase, and cool-down.

Different sociodemographic, cognitive, and physical condition variables will be evaluated. All dependent variables will be measured before and after the intervention, and statistical analysis will determine which exercise prescription yielded the best results in terms of cognitive improvement. This research aims to provide valuable information about the optimal dose of high-intensity exercise to improve cognition in older adults with mild cognitive impairment in Colombia."

DETAILED DESCRIPTION:
This research corresponds to an experimental study, a randomized single-blind controlled clinical trial, in which a total of 118 individuals, both men and women aged over 65, will participate. They will be divided into four groups: the control group (n = 31) and three experimental groups (n = 29 each). The variables will be measured for both groups using the same validated tools and evaluated by the same assessor to prevent information biases and differential misclassification. Evaluations will occur at the start of the intervention and immediately after its completion, with the results recorded in a data log. Subsequently, these results will be consolidated into an Excel database, with each participant assigned a code to ensure privacy while allowing for the necessary comparability.

Regarding the independent variables, we will address sociodemographic characteristics, clinical history, and the socio-familial assessment scale. As for the outcome variables, they are categorized into several areas: those related to health status will assess the relative risk of death due to comorbidity using the Charlson Comorbidity Index, health-related quality of life using the SF36 questionnaire, and Fried's frailty phenotype. Physical condition variables will be evaluated using the Senior Fitness Battery, gait and balance using the Tinetti Scale, and gait speed with the 6-minute walk test. Functional variables will be assessed using the Katz Index (activities of daily living), the Lawton & Brody Index (instrumental activities of daily living), and Siu and Reuben's Physical Scale (advanced activities of daily living). For the cognitive variable, we will employ the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA). Attention and executive functions will be measured using the Trail Making Test Part A and Part B. Verbal fluency will be assessed with the Verbal Fluency Test (VFT), while selective attention and concentration will be evaluated using the D2 test. Processing speed will be determined through the Digit Symbol Substitution Test (DSST).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 65 who voluntarily agree to participate in the study and are not engaged in any other physical exercise program
* Possess adequate physical autonomy to participate in the required physical activities for the study
* Exhibit mild cognitive impairment (with a score of <25 on the Mini-Mental State Examination)
* Have the capacity to comprehend the instructions, programs, and protocols of this trial.

Exclusion Criteria:

* People with contraindications for physical or exercise tests will be excluded. This includes individuals diagnosed with pathologies such as cancer, pulmonary hypertension, renal failure, heart failure, orphan diseases, psychiatric conditions, neurological or cognitive impairments, or Human Immunodeficiency Virus (HIV/AIDS) infection or disease.
* Individuals who do not consent to participate in the study or have declined to endorse the use of their data for research purposes in the informed consent at the time of program entry will also be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
General cognition | Up to twelve weeks
  General cognition will be assessed with the Montreal Cognitive Assessment (MoCA), which evaluates executive and visuospatial function, memory, attention, language, abstraction, recall memory, and orientation. The total possible score is 30 points; a score of 26 or above is considered normal.
Senior Fitness Battery (SFB) | Up to twelve weeks
  Physical condition and functional capacity variables will be assessed using the Senior Fitness Battery (SFB). The SFB includes tests for upper and lower limb muscle strength (arm curl and chair stand tests, respectively), aerobic capacity (6-minute walk test), lower limb flexibility (sit-and-reach test), upper limb flexibility (back scratch test), and dynamic agility and balance (8-foot up-and-go test).

SECONDARY OUTCOMES:
Trail Making Test part A and part B | Up to twelve weeks
  Attention and executive functions will be evaluated using the Trail Making Test part A and part B (TMTA and TMTB, respectively). These tests involve timed visual and motor tasks where participants must connect numbered circles consecutively (TMTA) or alternate circles of numbers and letters (TMTB). TMTA assesses psychomotor attention and speed, as well as the ability to switch between different tasks or rule sets, while TMTB assesses executive function. A shorter time to connect all circles is indicative of better attention and executive function. An average score for TMT-A is 29 seconds and a deficient score is greater than 78 seconds. For TMT-B, an average score is 75 seconds and a deficient score is greater than 273 seconds.

OTHER OUTCOMES:
Verbal fluency | Up to twelve weeks
  Verbal fluency will be assessed using the Verbal Fluency Test (VFT), widely used in neuropsychological assessments. Participants are asked to name as many animals as possible in one minute, without using higher categories like "fish" or lower categories. A score of under 17 indicates concern.
D2 test | Up to twelve weeks
  Selective attention and concentration will be evaluated with the D2 test. Selective attention focuses on the subject's ability to quickly discriminate and select a specific visual stimulus (e.g., the letter "d" with two marks) among other distracting stimuli that appear randomly. This time-limited test assesses the ability to follow instructions and discriminate stimuli, with scores divided into total correct, error percentage, total test efficiency calculated from the difference between processed words and errors, and a concentration index obtained from the difference between total correct and commission errors.
Digit Symbol Substitution Test (DSST) | Up to twelve weeks
  Processing speed will be evaluated using the Digit Symbol Substitution Test (DSST), a paper-and-pencil cognitive test that requires the subject to relate symbols to numbers according to a key located at the top of the page. The subject copies the symbol in spaces below a row of numbers. The score is based on the number of correct symbols within the allotted time, typically 90 to 120 seconds, with a maximum score of 60.
Tinetti scale | Up to twelve weeks
  The Tinetti scale evaluates postural stability, balance, and gait to determine a patient's risk of falls. The assessment is divided into two parts: the first assesses balance, with a maximum score of 16, and the second assesses gait, with a maximum score of 12. The total score, obtained by summing both parts, is used to classify fall risk.
Frailty phenotype | Up to twelve weeks
  Frailty was assessed using the frailty phenotype, consisting of five criteria: (i) involuntary weight loss; (ii) self-reported exhaustion; (iii) slow walking speed; (iv) weakness; and (v) low physical activity. An older adult with >3 criteria was classified as frail, while those with only 1 or 2 criteria were classified as moderately frail, and those with no criteria were classified as non-frail.
Katz index | Up to twelve weeks
  The Katz Index examines activities of daily living (ADLs) such as bathing, dressing, toileting, transferring, continence, and feeding, considering the dependence or independence in performing these activities. It was designed for use in individuals over 65 years of age and has been validated for universal applicability. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Lawton and Brody Index | Up to twelve weeks
  The Lawton and Brody Index evaluates instrumental activities of daily living (IADLs) such as shopping, cooking, cleaning, laundering, finances, medication, transportation, and phone use. It considers instrumental disability as the inability to perform one or more activities and has been validated in Spanish for the geriatric population. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
Siu and Reuben Physical Scale | Up to twelve weeks
  The Siu and Reuben Physical Scale for Advanced Activities of Daily Living (AADL) assesses the degree of integration and social relationships in older adults. This scale consists of 9 items, where each item is scored based on the time it takes the subject to perform the action. The scale has a maximum of 36 points, classifying the adult as autonomous (≥25) or non-autonomous (<25).

CONTACTS AND LOCATIONS:
Locations (1):
- Retos Salud Mental, Cali, Valle del Cauca Department, Colombia